CLINICAL TRIAL: NCT06756178
Title: Effect of Remimazolam Versus Dexmedetomidine on the Incidence of Delirium After Elective Cardiac Surgery with Cardiopulmonary Bypass: a Prospective Randomized Controlled Trial
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moataz Emad Eldin Omar Mohamed, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Elective cardiac surgery
Record Dates: First submitted 2024-12-17; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-11

CONDITIONS: Delirium - Postoperative
Keywords: cradiac surgery with cardiopulmonary bypass
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: Effect of Remimazolam versus Dexmedetomidine on the incidence of delirium post elective cardiac suregery
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 : propofol group (Placebo Comparator): Postoperative Use
  Interventions: Drug: Propofol Group 1
- Group 2: Remimazolam Intervention (Experimental): Postoperative Use
  Interventions: Drug: Remimazolam Intervention
- Group 3: Dexmedetomidine Intervention (Experimental): Postoperative Use
  Interventions: Drug: Dexmedetomidine Intervention

INTERVENTIONS:
Drug: Propofol Group 1 — Postoperative Use:
  Bolus: 10-20 mg intravenously as needed for sedation initiation. Continuous infusion: 0.3-0.5 mg/kg/hour to maintain light sedation adjusted based on clinical response.
  Arms: Group 1 : propofol group
Drug: Remimazolam Intervention — Postoperative Use:
  Initial bolus: 5 mg intravenously upon ICU arrival. Continuous infusion: 0.2-0.3 mg/kg/hour to maintain light sedation with a maximum dose of 0.8 mg/kg/hour.
  Rescue sedation with propofol or midazolam will be allowed if patients become agitated or if Remimazolam is ineffective in maintaining target sedation.
  Arms: Group 2: Remimazolam Intervention
Drug: Dexmedetomidine Intervention — Postoperative Use:
  Loading dose: 0.5-1 μg/kg over 10-20 minutes after ICU arrival. Continuous infusion: 0.2-0.7 μg/kg/hour for sedation maintenance, adjusted as needed to maintain light sedation.
  Rescue sedation with propofol or midazolam will be administered if Dexmedetomidine fails to maintain adequate sedation or if patients become agitated.
  Arms: Group 3: Dexmedetomidine Intervention

SUMMARY:
The study aims to improve the post-open heart surgery lifestyle and overall experience, as well as assess the incidence of delirium using Remimazolam and Dexmedetomidine.

DETAILED DESCRIPTION:
Delirium is an acute brain dysfunction characterized by an acute onset and fluctuating course of disturbance in attention, awareness, and cognition, It is the most common neurocognitive complication following cardiac surgery, with an incidence rate between 11% and 52%.

The occurrence of delirium correlates strongly with various short- and long-term poor outcomes following cardiac surgery, including prolonged ICU stay and hospitalization and increased risk of hospital readmission. Different risk factors contribute to delirium after cardiac surgery, including advanced age, pre-existing cognitive impairment, diabetes, history of stroke, type of surgery, extended CPB duration, and blood transfusion. Dexmedetomidine is a highly and potently selective α2-adrenoceptor agonist with anxiolytic, sedative, and analgesic properties. It has neuroprotective effects by reducing neuroinflammation, apoptosis, and blood-brain barrier injury via central α2A adrenoceptors, but it can cause hypotension and bradycardia.

Remimazolam, a new ultra-short-acting benzodiazepine, also has a faster onset of action and a higher safety profile. It was recently approved for procedural sedation and general anesthesia. Its metabolism is mainly induced by tissue esterase, independent of liver and kidney function, and its metabolites are inactive. In addition, flumazenil reverses the effects of Remimazolam in the event of adverse events, an advantage not available in non-benzodiazepines. The objective of this clinical trial is to evaluate the efficacy of Remimazolam compared with Dexmedetomidine for preventing postoperative delirium after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Scheduled for cardiac surgery (CABG and/or valve replacement).
* Elective surgery

Exclusion Criteria:

* Patients with known allergies to Remimazolam or Dexmedetomidine
* Refusal to participate.
* History of psychiatric or neurological conditions (schizophrenia, epilepsy, severe dementia, etc.).
* Preoperative inability to communicate (severe visual/auditory dysfunction, language barriers).
* Severe hepatic or renal dysfunction
* Cardiopulmonary bypass time not ≥ 120 minutes
* aortic clamping time not ≥ 90 minutes
* Emergency surgeries
* On preoperative mechanical ventilation and long sedation time
* reoperated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Delirium (POD) | During the first 5 days after surgery
  Delirium will be assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) twice daily during the first 5 days after surgery

SECONDARY OUTCOMES:
Time of delirium onset and duration ,Sedation level | During first 5 days after surgery
  1. Time of delirium onset and duration until the end of it.
  2. Sedation level: Assessed using the Richmond Agitation-Sedation Scale (RASS).

OTHER OUTCOMES:
ICU length of stay ,Length of Stay in Hospital After Surgery | From end of surgery until discharge from Intensive Care Unit or 30 days after surgery. From end of surgery until discharge from hospital or 30 days after surgery
  Results will be presented as median (95% confidence interval)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The effect of perioperative dexmedetomidine on postoperative delirium in adult patients undergoing cardiac surgery with cardiopulmonary bypass — https://link.springer.com/article/10.1186/s12871-024-02715-2
- See also: Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine — https://link.springer.com/article/10.1007/s40262-017-0507-7
- See also: The neuroprotective effect of dexmedetomidine and its mechanism — https://www.frontiersin.org/journals/pharmacology/articles/10.3389/fphar.2022.965661/full
- See also: Remimazolam: First Approval — https://link.springer.com/article/10.1007/s40265-020-01299-8
- See also: Remimazolam besilate, a benzodiazepine, has been approved for general anesthesia — https://link.springer.com/article/10.1007/s00540-020-02755-1